CLINICAL TRIAL: NCT07258797
Title: Short Course or Long Course Radiotherapy as Total Neoadjuvant Therapy in Locally Advanced Rectal Cancer : A Prospective, Open Label, Single Institution, Randomized, Parallel Arm Comparative Study
Brief Title: Short Course or Long Course Radiotherapy as Total Neoadjuvant Therapy in Locally Advanced Rectal Cancer
Acronym: SHOOL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Shaifali Goel, Consultant, Department of Gastrointestinal and Hepatobiliary services, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGCIRC/IRB-BHR/52/2025
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Adenocarcinoma of the Rectum
Keywords: SHORT COURSE RADIOTHERAPY; LONG COURSE RADIOTHERAPY; RECTAL CANCER; OUTCOMES; SURVIVAL
MeSH Terms: conditions — Rectal Neoplasms | interventions — Consolidation Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCRT + Consolidation Chemotherapy (Active Comparator): Radiotherapy: 25 Gy in 5 fractions over 1 week to the pelvis using IGRT technique.
  1. Interval before Chemotherapy: 1-2 weeks after completion of radiotherapy.
  2. Chemotherapy: Modified FOLFOX6 every 2 weeks (total of 12 cycles).
  Interventions: Radiation: SCRT : 25 Gy in 5 fractions over 1 week to the pelvis using IGRT technique
- LCRT + Consolidation Chemotherapy (Active Comparator): Radiotherapy:
  1. Primary tumor and involved nodes: 50 Gy in 25 fractions.
  2. Elective nodal basin: 45 Gy in 25 fractions. Delivered concurrently with oral Capecitabine (825 mg/m² twice daily on radiotherapy days).
  Interventions: Radiation: LCRT + Consolidation Chemotherapy

INTERVENTIONS:
Radiation: SCRT : 25 Gy in 5 fractions over 1 week to the pelvis using IGRT technique — Arm A - SCRT + Consolidation Chemotherapy
  1. Radiotherapy: 25 Gy in 5 fractions over 1 week to the pelvis using IGRT technique.
  2. Interval before Chemotherapy: 1-2 weeks after completion of radiotherapy.
  3. Chemotherapy: Modified FOLFOX6 every 2 weeks (total of 12 cycles). If the patient is fit, the option of intensifying the chemo to mFOLFIRINOX will be discussed with the patient
  Arms: SCRT + Consolidation Chemotherapy
Radiation: LCRT + Consolidation Chemotherapy — Arm B - LCRT + Consolidation Chemotherapy 1) Radiotherapy: o Primary tumor and involved nodes: 50 Gy in 25 fractions. o Elective nodal basin: 45 Gy in 25 fractions. Delivered concurrently with oral Capecitabine (825 mg/m² twice daily on radiotherapy days). o Technique: IGRT 2) Interval before Chemotherapy: 1-2 weeks after completion of chemoradiotherapy. 3) Chemotherapy: Modified FOLFOX6
  Arms: LCRT + Consolidation Chemotherapy

SUMMARY:
This study compares two standard radiotherapy approaches (short-course vs. long-course) given before surgery in patients with locally advanced rectal cancer. The goal is to see which treatment is more effective and better tolerated.

DETAILED DESCRIPTION:
The SHOOL study is a single-institution, open-label, randomized prospective study designed to evaluate and compare two internationally accepted total neoadjuvant therapy (TNT) strategies in patients with locally advanced rectal cancer (LARC). These strategies differ primarily in their radiotherapy schedule and include:

Arm A: Short-course radiotherapy (SCRT; 25 Gy in 5 fractions over 1 week), followed by consolidation chemotherapy and surgery

Arm B: Long-course chemoradiotherapy (LCRT; 50.4 Gy in 28 fractions with concurrent Capecitabine over 5-5.5 weeks), followed by consolidation chemotherapy and surgery The study acronym "SHOOL" reflects the clinical dilemma of whether SHOrt-course Or Long-course radiotherapy offers better or more practical outcomes when delivered within a TNT framework.

This prospective study aims to explore how these two strategies compare in terms of tumour response (as measured by pathological complete response, pCR), toxicity, treatment compliance, feasibility, quality of life, and local recurrence rates at 3 and 5 years. Given that both arms represent evolving standards of care, this study is designed to generate real-world data that can guide institutional decision-making and inform future definitive trials.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the rectum
2. Locally advanced disease based on MRI including cT3-T4 and/or node positive disease (cN1 or N2)
3. Tumor located within 15 cm from the anal verge (confirmed by endoscopy or MRI)
4. ECOG performance status 0-2
5. Hemoglobin ≥ 9 g/dL
6. Absolute neutrophil count ≥ 1,500/mm³
7. Platelets ≥ 100,000/mm³
8. Total bilirubin ≤ 1.5 × ULN
9. Aspartate transaminase/Alanine transaminase ≤ 2.5 × ULN
10. Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min
11. Fit for neoadjuvant therapy and curative resection
12. Willing and able to provide written, informed consent
13. Baseline MRI and biopsy (even if done outside) must be reviewed and approved by the institutional radiology and pathology review board, requiring concurrence from two independent pathologists and two independent radiologists

Exclusion Criteria:

1. Metastatic disease at presentation (distant nodes, liver, lung, peritoneum, etc.)
2. Prior pelvic radiotherapy or systemic chemotherapy for rectal cancer
3. Presence of synchronous malignancies or previous malignancy within 5 years except: Treated basal cell or squamous cell carcinoma of the skin, In situ cervical cancer, Active uncontrolled infection
4. Known HIV infection with CD4 < 200 cells/μL, or active hepatitis B or C
5. Severe comorbid conditions precluding therapy (e.g., decompensated cardiac, hepatic, or renal disease)
6. Pregnant or breastfeeding women
7. Inability to comply with protocol requirements or follow-up schedule
8. Psychiatric illness or social situations that may limit compliance with study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate measured in proportion of participants (%) | 3 and 5 years
  Proportion of participants achieving pathological complete response, defined as ypT0N0 on histopathological examination of resected tumor specimens after surgery. Assessment will be performed by institutional pathologists according to standardized reporting guidelines. The pCR rate is central to evaluating early tumor response to total neoadjuvant therapy.
  Unit of Measure:
  Proportion of participants (%)

SECONDARY OUTCOMES:
Local Recurrence Rate measured in percentage of participants (%) | 3 and 5 years
  Proportion of participants experiencing loco-regional relapse, defined as reappearance of tumor at the primary site or regional lymph nodes, as confirmed by clinical evaluation and imaging (pelvic MRI or CT scan) at specified intervals post-treatment.
  Unit of Measure:
  Percentage of participants (%)
Overall Survival (OS) in months | Evaluated at 3 years and 5 years
  Overall survival is defined as the time from randomization to death from any cause. Participants who are alive at the time of analysis or are lost to follow-up will be censored at the last date known to be alive. Outcome will be summarized using median survival and survival rates at specified time points.
  Unit of Measure:
  Time in months
Acute Toxicities graded using CTCAE version 5.0 | 3 months post surgery
  All adverse events occurring during RT and chemotherapy up to 3 months post-surgery
Late Toxicities documented using clinician assessment and patient reported outcomes EORTC QLQ-C30 and QLQ-CR29 | 6 months to 2 years post-treatment
  Number and proportion of participants experiencing treatment-related adverse effects arising between 6 months and 2 years post-treatment, including bowel dysfunction (e.g., frequency, urgency), bladder dysfunction (e.g., incontinence, retention), and sexual dysfunction. Assessment will be performed through standardized clinician evaluation and patient-reported outcome measures using validated questionnaires.
  Unit of Measure:
  Percentage of participants (%)
Treatment completion Rate measured in percentage of participants (%) | 1 year
  Proportion of participants who complete the planned treatment regimen, including radiotherapy (RT), chemotherapy cycles, and surgery. Reasons for any deviations from the planned treatment, such as toxicity, patient refusal, or disease progression, will be documented and analyzed.
  Unit of Measure:
  Percentage of participants (%)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 1 year
  Assessed by the proportion of participants adhering to the treatment protocol as planned, rates of treatment delays or dose reductions due to adverse events, and multidisciplinary team (MDT) decision-making trends regarding treatment modifications. These measures collectively evaluate the practical implementation and patient tolerance of the therapeutic regimen.
  Unit of Measure:
  Percentage of participants (%) and descriptive trends

CONTACTS AND LOCATIONS:
Overall Officials: Jaskaran Sethi, MD, Study Director — Rajiv Gandhi Cancer Hospital and Research Centre, New Delhi
Locations (1):
- Rajiv Gandhi Cancer Institute and Research Centre, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified data sets will include participant demographics, baseline measures, intervention details, clinical outcomes, and adverse events recorded during the study.
Supporting Information: Study Protocol, ICF
Time Frame: IPD and supporting information will be available beginning six months after publication of the primary results or completion of the study, whichever is later. Data will remain accessible for five years from the start date of availability.
Access Criteria: Qualified researchers who submit a methodologically sound research proposal will be able to access de-identified individual participant data underlying the main results, as well as supporting documents such as the study protocol and statistical analysis plan. Access will be granted through a secure data sharing portal, subject to data use agreements that ensure participant confidentiality and limit use to the specified research purpose

REFERENCES:
- [Background] Bahadoer RR, Dijkstra EA, van Etten B, Marijnen CAM, Putter H, Kranenbarg EM, Roodvoets AGH, Nagtegaal ID, Beets-Tan RGH, Blomqvist LK, Fokstuen T, Ten Tije AJ, Capdevila J, Hendriks MP, Edhemovic I, Cervantes A, Nilsson PJ, Glimelius B, van de Velde CJH, Hospers GAP; RAPIDO collaborative investigators. Short-course radiotherapy followed by chemotherapy before total mesorectal excision (TME) versus preoperative chemoradiotherapy, TME, and optional adjuvant chemotherapy in locally advanced rectal cancer (RAPIDO): a randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Jan;22(1):29-42. doi: 10.1016/S1470-2045(20)30555-6. Epub 2020 Dec 7. PMID 33301740